CLINICAL TRIAL: NCT06605729
Title: Physio Perspective Study
Brief Title: Exploring Physiotherapist's Knowledge, Attitudes, Beliefs and Clinical Decision-making Regarding Physical Activity in Chronic Pain Management.
Acronym: PPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Prof. dr. Mira Meeús, Prof. dr. Mira Meeus, Universiteit Antwerpen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: B3002022000133; Project ID 3805 (Other: University of Antwerp)
Record Dates: First submitted 2024-09-04; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Cancer Survivorship; Chronic Low Back Pain (CLBP); Physiotherapy and Rehabilitation
Keywords: Physiotherapy and rehabilitation; Clinical Decision Making; Attitudes and beliefs; Physical Activity; Chronic Pain; Cancer Survivorship; Knowledge; Chronic Low Back Pain; elearning
MeSH Terms: conditions — Behavior; Motor Activity; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- e-learning (Experimental): The aim of the educational module intervention is to enhance the knowledge, attitudes, beliefs and behavior of HCPs about physical activity as a part of the management of chronic pain. The content of is based on most recent scientific knowledge and guidelines about the management of chronic pain and physical activity and on behavioral change. Four themes are presented: chronic pain, physical activity and chronic pain, specific populations and behavior change.
  Each subpart can be studied separately. Having separated chapters will be easier for participants to navigate the content, to follow along and to be able to integrate the knowledge in their daily practice. The module will be available online through Teachable™ and will contain a mixture of video and additional written material. Completing the complete module will take approximately 2 hours.
  Interventions: Other: e-learning

INTERVENTIONS:
Other: e-learning — The content of this e-learning is based on most recent scientific knowledge and guidelines about the management of chronic pain and physical activity and on behavioral change. Four themes are presented: chronic pain, physical activity and chronic pain, specific populations and behavior change.

SUMMARY:
Chronic pain is a globally increasing problem, with enormous impact on the individual and society. Within the treatment of chronic pain, physical activity is a key strategy to improve pain-related complaints. There is ample evidence that physical activity has numerous benefits and few drawbacks. However, the literature shows that those who experience chronic pain experience difficulty performing and sustaining physical activity, and several barriers emerge that hinder physical activity. Patients indicate a need for the supportive role of the health care provider when it comes to guidance toward physically active lifestyle. On the other hand, caregivers find it difficult to fill this role. This can cause frustration for both parties, with a negative impact on the delivery of care.

Within the treatment of chronic pain, the physiotherapist is an important healthcare provider. However, it is currently not clear how physiotherapists fulfill their role in the treatment of a patient with chronic pain. It is also not known what the current knowledge is among physiotherapists on chronic pain management, what the perceptions and beliefs around physical activity in the treatment of chronic pain are, and what the clinical decisions are that they make in the treatment of chronic pain in terms of physical activity.

To obtain the best and broadest possible answers to these research questions, this study will examine these themes among physiotherapists with respect to two patient groups; namely, patients who experience persistent pain after completing their cancer treatment and individuals with chronic low back pain.

Demographic data such as age, employment, occupational specializations, etc. is gathered. Furthermore, knowledge of chronic pain, underlying thoughts and perceptions around chronic pain and physical activity, and clinical decisions of a physiotherapist in treating a patient with chronic pain, including decisions about physical activity will be examined.

In addition, this study also investigates whether an elearning around chronic pain and physical activity, has an effect on these knowledge and treatment actions.

Participants will be asked to complete a set of questionnaires at 2 time points via an online platform. A first measurement moment happens at the start of the study, after this the participant gets access to the elearning, the second measurement moment happens 30 days after the first measurement moment.

DETAILED DESCRIPTION:
Pain is one of the most common, complex and persisting symptoms worldwide. Next to the debilitating impact on the individual, pain also has a social and economic impact. A classification of pain based on duration provides the distinction between acute and chronic pain, with chronic pain described as persistent or recurrent pain for at least 3 months. The chronic pain population consists of patients with a broad variety of medical conditions. In the literature, a discrimination based on the associated condition is often made, with the most frequent distinction between non-cancer and cancer-related pain. Cancer-related pain is a debilitating symptom with a pain prevalence of 39.3% after curative cancer treatment. Within the non-cancer related pain, spinal pain has the highest prevalence and low back pain leads the chart of the years with lived disability.

Despite the different underlying condition, physical activity and exercise are the main part of the best-evidence treatment for chronic pain, both in the population of cancer survivors with chronic pain as well as in a population of chronic low back pain patients.

It is evident that this effectiveness cannot be attained without a long-term engagement towards physical activity and exercise behavior. Unfortunately, patient' adherence towards physical activity is low, which is a problem in most exercise interventions in the population under study. So, despite the benefits of physical activity for chronic pain, low physical activity levels are still reported across the span of these two populations.

Undertaking physical activity is a complex behavior with many aspects that need to be considered. Knowledge from qualitative studies clarify the self-reported barriers and facilitators towards physical activity that patients experience. This reveals similarities between experienced barriers and facilitators in patients from both populations. At a personal level it is seen that barriers on a physical level such as pain and barriers and on a psychological level such as low self-efficacy, are similar. What is also striking is that the health care provider (HCP) also has an important role to play in physical activity and exercise behavior. Uncertainty, a lack of clear information is experienced as a barrier and subsequently the need of supervision and support from an HCP is considered to be a facilitator. Additionally, previous evidence has already shown the influence of beliefs of HCPs on the beliefs of patients .

The experience of the patient shows that the HCP is part of the key in motivating towards exercise behavior. Yet, the current research on physical activity and exercise behavior of patients with chronic pain lacks the perspective of the HCP. It is known that HCPs with a biomedical view prescribe less active treatment strategies and more advice to rest in chronic low back pain patients. However, most research on physical activity prescription behavior stays quite general and therefore, it is not known what exactly they do or don't prescribe. Next to that, it is unclear what the beliefs and attitudes are of the HCPs towards physical activity and exercise in chronic pain management and how that determines this prescription behavior. A group of HCPs who are likely to prescribe and use exercise in their treatment are physiotherapists. In line with research on other HCPs, it remains unclear how physiotherapists actually recommend and organize physical activity for their patients with chronic pain. Additionally, it is not known whether the manner wherein they prescribe physical activity might differ based on their biomedical or biopsychosocial orientation, on their beliefs of the associated condition and on the beliefs on physical activity in relation to chronic pain. This knowledge will help to understand the physical activity and exercise prescription of physiotherapists and clarify how this might influence physical activity levels in the patient population of chronic pain, more specifically chronic low back pain patients and cancer survivors with chronic pain. The inclusion of these two population-groups, both with varied challenges, offers an opportunity to increase the generalizability of these findings across chronic pain conditions and to obtain broad insights into the experiences of people with chronic pain.

Gaining more insight in the behavior, the beliefs about and attitudes towards physical activity in physiotherapists who work with chronic pain patients is the first piece of the puzzle in better supporting patients with chronic pain in their physical activity journey.

Thereforen, this study has three objectives:

1. To explore the knowledge, the attitudes and beliefs, and the clinical decision making in chronic pain management, including physical activity as part of this management of physiotherapists with clinical expertise in:

   * chronic low back pain.
   * chronic pain in cancer survivorship.
2. To compare the knowledge, the attitudes and beliefs, and the clinical decision making in chronic pain management between these two groups.
3. To research if an eLearning can change knowledge, the attitudes and beliefs, and the clinical decision making in chronic pain management, including physical activity as part of this management of physiotherapists with clinical expertise in:

   * chronic low back pain.
   * chronic pain in cancer survivorship.

This is a uncontrolled clinical trial study design. Physiotherapists interested in the study will be invited to connect to the online platform and read the informed consent about the study.

The study will be conducted through an online survey, consisting of questionnaires and a clinical case with questions. Following data will be collected through the survey:

1. Demographic data.
2. Knowledge on chronic pain.
3. Implicit and explicit beliefs and attitudes on chronic pain management, including physical activity as part of pain management.
4. Clinical decision making in chronic pain management, including decisions on physical activity.

Baseline assessment is completed in one sitting and is estimated to last 30 minutes. After finishing this first part, they will be invited for an eLearning. The educational module consists of video-material, implementation exercises and additional literature. Each participant has an individual login on a protected digital platform from which content cannot be downloaded or shared, and will be able to access the module for 30 days.

After 30 days, each participant will be asked to repeat the same questionnaires, regardless if they completed the module or not.

ELIGIBILITY:
Inclusion Criteria:

* To be able to read and write Dutch.
* To have access to a computer with an internet connection.
* Currently working as a physiotherapist in Belgium or the Netherlands.
* Experience with the population at hand.

Exclusion Criteria:

* currently not working as a physiotherapist.
* Other health care professionals.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
KNAP | At baseline and at 30 days
  The Dutch Knowledge and Attitude on Pain (KNAP) questionnaire will be administered. It is a 30-item questionnaire which measures the knowledge on chronic pain and pain neurophysiology, biomedical or biopsychosocial beliefs on chronic pain and explicit beliefs on pain management strategies, including physical activity. Questions are statements that are scored on a 6 point Likert-scale, that ranges between: totally not agree (1) and totally agree (6). The total score ranges from 30-180, where a higher overall score indicates better knowledge on pain neurophysiology and a more modern pain-management approach. The KNAP has good measurement properties to evaluate HCPs' knowledge on and attitudes towards modern pain neuroscience.

SECONDARY OUTCOMES:
Clinical Case Questionnaire | At baseline and at 30 days
  A clinical case of a patient of the population of interest (chronic low back pain patient or a cancer survivor with chronic pain) will be presented. Questions on clinical reasoning, on physical activity guideline knowledge and on clinical decisions regarding treatment and physical activity prescription behavior for this specific patient provide quantitative and qualitative data through open, closed and Likert-scale questions on clinical decision making on the treatment plan in general and specific questions on physical activity and exercise prescription. Based on the answers to the questionnaire, physical activity prescription behaviour will be categorized into different categories: choice of level of intensity, choice of used body part, choice to load or deload the painful area, guideline adherent or not. There is no total score and results of this questionnaire are descriptive in nature.
IAT | At baseline.
  An implicit association task (IAT) is a test to counter the bias of social desirability in measuring beliefs and attitudes. In these tests, the participant needs to rapidly categorize two target concepts (in this study: "Rest" and "Activity") with an attribute (in this study: "Safe" or "Dangerous"). The IAT rests on the assumption that it is easier to make the same behavioral response (pressing a key on a keyboard) to concepts that are strongly associated than to concepts that are weakly associated. The faster response indicates an easier pairing of the concept and attribute, which means that this association is stronger than the slower response association. The outcome of an IAT is the response time to each combination of target concepts and attributes where a short response time indicates a strong association and a longer time a weak association.

CONTACTS AND LOCATIONS:
Overall Officials: Mira Meeus, Doctoral degree, Principal Investigator — Universiteit Antwerpen; Nathalie Roussel, Doctoral degree, Study Chair — Universiteit Antwerpen; An De Groef, Doctoral degree, Study Chair — Universiteit Antwerpen
Locations (1):
- University of Antwerp, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided